CLINICAL TRIAL: NCT02336035
Title: Unstable Distal Radius Fractures in Patients Over 65 Years. Conservative Treatment With Cast Immobilization Versus Volar Locking Plate. A Prospective Randomized Controlled Trial.
Brief Title: Distal Radius Fractures in Patients Over 65 Years, Operation or Cast?
Acronym: DROC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sondre Stafsne Hassellund, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014 3830 RCT radius 65
Record Dates: First submitted 2015-01-05; First posted 2015-01-12 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cast immobilization (No Intervention): Cast immobilization for 5 weeks from primary injury/reduction. Thereafter active exercise within the range of pain.
  Both groups will be followed after 3, 6 and 12 months, and after 2 and 5 years.
- Operation (Experimental): Operation with a volar plate. Cast immobilization for 2 weeks after operation, thereafter active motion without weight for 4 weeks. 6 weeks after operation the patients are allowed active exercise within the range of pain.
  Both groups will be followed after 3, 6 and 12 months, and after 2 and 5 years.
  Interventions: Procedure: Volar plate

INTERVENTIONS:
Procedure: Volar plate — Flexor carpi radialis (FCR)-approach. Standard surgical procedure with a volar locking plate
  Other Names: Volar locking plate; VLP
  Arms: Operation

SUMMARY:
Eligible patients that sign an informed consent will be randomized to operation with volar locking plate or cast immobilization. Primary follow-up after 1 year.

DETAILED DESCRIPTION:
The investigators want to investigate if there is a difference between operative treatment with volar locking plates and cast immobilization in patient above 65 years with unstable distal radius fractures AO/OTA type A and C . Eligible patients that meets the radiological criteria (see inclusion criteria) will be randomized to cast immobilization or operation with volar locking plate.

The investigators are planning a non-inferiority design.

The current study will test the following null hypothesis:

In patients over 65 years of age with unstable distal radius fractures AO/OTA type A and C,volar locking plates are superior to cast immobilization by more than 8 points, as evaluated by quick-DASH at 12 months follow-up.

The investigators will perform a cost-effectiveness analysis comparing QALYs (Quality-adjusted life years) and costs with the two interventions the first year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* AO/OTA class A- and C-fractures
* Age > 65 years
* Unacceptable primary reduction or redislocation < 20 days post-injury with at least one of the following findings:
* dorsal angulation > 10 degrees
* radial shortening > 3 mm
* intraarticular step-off > 2 mm
* Ability to sign an informed consent
* Acute fracture, inclusion within 20 days from injury.
* Ability to reconstruct the articular surface with a volar locking plate

Exclusion Criteria:

* Volar angulated fractures and AO type B
* Associated diseases contraindicating surgery
* Mental impairment, nursery home patient
* Earlier wrist injury
* Pathological fractures
* Open fractures (>Gustilo-Anderson I) or damaged soft tissue
* Drug abuse
* Concomitant injuries that might affect outcome
* Congenital anomaly of affected extremity
* Median nerve compression that requires acute operation
* Foreign language
* Tourists

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-09 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Quick disabilities of the arm, shoulder and hand; Quick-DASH | 1 year
  Questionnaire

SECONDARY OUTCOMES:
Quick DASH | 3 and 6 months; 2 and 5 years
  Questionnaire
Patient rated wrist evaluation (PRWE) | 3, 6 and 12 months; 2 and 5 years
  PRWE, Questionnaire
Grip strength | 3, 6 and 12 months; 2 and 5 years
  score
Range of motion | 3, 6 and 12 months; 2 and 5 years
  score
Over all satisfaction | 6 weeks; 3, 6 and 12 months; 2 and 5 years
  Over all satisfaction with hand function, numeric scale 0-10
Complications | 6 weeks; 3, 6 and 12 months; 2 and 5 years
  Registration of complications
X-ray, wrist | 6 weeks; 3 and 12 months; 2 and 5 years
  Radial shortening, dorsal tilt, intraarticular step-off
EQ-5d (EuroQol) | 6 weeks; 3, 6 and 12 months; 2 and 5 years
  Questionnaire
Registration of need for assistance in daily life | 6 weeks; 3, 6 and 12 months; 2 and 5 years
  Registration of need for assistance in daily life to register costs generated

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Madsen, Professor, Study Chair — University of Oslo
Locations (1):
- Oslo University hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided